CLINICAL TRIAL: NCT04649372
Title: EndoVE endosCopic Treatment for Oesophageal and Gastric canceR
Acronym: VECTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mirai Medical (Industry)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-20-001(MM-CC-100)
Record Dates: First submitted 2020-11-18; First posted 2020-12-02 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2021-01

CONDITIONS: Oesophageal Cancer; Oesophageal Disease; Gastric Cancer
Keywords: Palliation
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoVE endosCopic Treatment for Oesophageal and Gastric canceR (Other): The patient will be placed under General Anaesthetic or sedated before Bleomycin will be delivered intravenously. The patient will then be treated endoscopically with the EndoVE device. The EndoVE procedure should take no longer than 30 minutes. The patient will then be transferred to the step-down ward to monitor for any adverse events before being discharged. There will be a telephone follow up after 2 days, 7 days, 4 weeks and 8 weeks. The patient will be requested to attend the clinic for a 12-week follow up for clinical review.
  Interventions: Procedure: EndoVE

INTERVENTIONS:
Procedure: EndoVE — On the day of the procedure, a review of any changes which occurred since the pre-study visit will be conducted. The patient will be placed under general anaesthesia or sedated before Bleomycin will be delivered intravenously. The patient will then be treated endoscopically with the EndoVE device. The EndoVE procedure should take no longer than 30 minutes.
  Other Names: ePORE

SUMMARY:
This project aims to establish the safety and efficacy of treating patients with inoperable oesophageal cancer or gastric cancer, using an endoscopic electroporation system (EndoVE) to facilitate direct chemotherapy tumour absorption.

DETAILED DESCRIPTION:
The use of electroporation has expanded over the last twenty years since its first clinically reported study in the treatment of head and neck cancer in 1991.

In electroporation short high-voltage pulses are delivered directly to the tumour which transiently permeabilises the cell membranes enabling targeted cell death and also allowing otherwise non-permeant chemotherapeutic drugs to enter the cancer cells. The parameters of a successful electroporation process are determined by the strength of the electric field and the duration of the electrical field exposure. ePORE and EndoVE deliver electroporation parameters which successfully electroporate cells in the reversible electroporation range, whilst eliminating muscular contractions. Both devices are CE marked and will be used within the definition of their intended use.

Currently over 150 sites in Europe are reported to be employing electroporation in the clinical management of head & neck, recurrent breast, malignant melanoma, colorectal, liver metastasis, pancreatic and inoperable glioma. The standard operating procedures for electroporation and electrochemotherapy were established during the EU funded ESOPE study which established the clinical application of electroporation in combination with cisplatin or bleomycin. The EndoVE device has already been used successfully in phase I studies in patients with inoperable oesophageal and colorectal cancer. No serious adverse events were noted with positive tumour regression observed after a single treatment.

A patient recruited to the study will be requested to attend a pre-study visit where informed consent will be obtained before proceeding to review medical history and conduct a full clinical examination, full blood count, EKG and assessment of tumour volume via a CT. The procedure will happen no later than 28 days after the pre-study visit - Day 0.

On the day of the procedure, a review of any changes which occurred since the pre-study visit will be conducted. The patient will be placed under General Anaesthetic or sedated before Bleomycin will be delivered intravenously. The patient will then be treated endoscopically with the EndoVE device. The EndoVE procedure should take no longer than 30 minutes. The patient will then be transferred to the step-down ward to monitor for any adverse events before being discharged. There will be a telephone follow up after 2 days, 7 days, 4 weeks and 8 weeks. The patient will be requested to attend the clinic for a 12-week follow up for clinical review,

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified oesophageal tumour
* Men or women aged at least 18 years of age.
* Patient has already received or been considered for surgery, and / or chemo-radiation.
* Performance status (Karnofsky > 60% or ECOG/WHO <2).
* Treatment free interval of at least 2 weeks after previously applied therapy.
* Patients must be mentally capable of understanding the information given.
* Patients must give written informed consent.

Exclusion Criteria:

* Coagulation disorder.
* Patients with a clinically manifested arrhythmia or with a pacemaker.
* Patients with oesophageal stenosis that cannot be relieved via balloon dilation.
* Oesophageal tumour treated with radiotherapy in the previous 4 weeks.
* Patients with epilepsy.
* Pregnancy or lactation/breastfeeding.
* Patients known to be Hepatitis B/C or HIV positive.
* Concurrent treatment with an investigational medicinal product or participation in another clinical study.
* Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
* Highly ulcerated oesophageal tissue.
* Contraindications for bleomycin use including acute pulmonary infection and severe pulmonary disease.
* Allergic reactions to bleomycin observed previously
* If a bleomycin cumulative dose of 400 x103 IU has been exceeded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (CTCAE) | 12 weeks
  Safety evaluation will be performed via continuous assessment of safety parameters by reviewing events as they arise. The investigation will be put on hold if unacceptable safety issues are outstanding.
  Adverse Events (AE) and Serious Adverse Events (SAE) will be evaluated and graded according to Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Efficacy of system in palliation of dysphagia | 12 weeks
  Change in dysphagia post treatment as measured by Ogilvie Dysphagia Score
Response Evaluation Criteria in Solid Tumours (RECIST) | 12 Weeks Post-Treatment
  Following CT scan at 12 weeks, a response evaluation will be conducted and reported.
Evaluation of Patient Reported Quality of Life (EORTC QLQ30) | Baseline (Day 0), Day 0 + 2 days, Day 0 + 1 week, Day 0 + 4 Weeks, Day 0 + 8 Weeks, Day 0 + 12 Weeks
  Change in Quality of Life Patient Reported Outcomes as measured by European Organisation for Research and Treatment of Cancer (EORTC) QLQ30
Evaluation of Patient Reported Quality of Life (EORTC QLQ-OES18) | Baseline (Day 0), Day 0 + 2 days, Day 0 + 1 week, Day 0 + 4 Weeks, Day 0 + 8 Weeks, Day 0 + 12 Weeks
  Change in Quality of Life Patient Reported Outcomes as measured by disease specific European Organisation for Research and Treatment of Cancer (EORTC) QLQ-OES18
Evaluation of Pain pre and post-treatment | Day 0 Pre-treatment, Day 0 Post-Treatment
  Change in pain experienced by the patient before and after treatment as measured by Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Simon Parsons, MD, FRCS, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jahangeer S, Forde P, Soden D, Hinchion J. Review of current thermal ablation treatment for lung cancer and the potential of electrochemotherapy as a means for treatment of lung tumours. Cancer Treat Rev. 2013 Dec;39(8):862-71. doi: 10.1016/j.ctrv.2013.03.007. Epub 2013 Apr 17. PMID 23601905
- [Background] Forde PF, Sadadcharam M, Bourke MG, Conway TA, Guerin SR, de Kruijf M, O'Sullivan GC, Impellizeri J, Clover AJP, Soden DM. Preclinical evaluation of an endoscopic electroporation system. Endoscopy. 2016 May;48(5):477-483. doi: 10.1055/s-0042-101343. Epub 2016 Apr 4. PMID 27042930
- [Result] Falk Hansen H, Bourke M, Stigaard T, Clover J, Buckley M, O'Riordain M, Winter DC, Hjorth Johannesen H, Hansen RH, Heeboll H, Forde P, Jakobsen HL, Larsen O, Rosenberg J, Soden D, Gehl J. Electrochemotherapy for colorectal cancer using endoscopic electroporation: a phase 1 clinical study. Endosc Int Open. 2020 Feb;8(2):E124-E132. doi: 10.1055/a-1027-6735. Epub 2020 Jan 22. PMID 32010744
- [Result] Egeland C, Baeksgaard L, Johannesen HH, Lofgren J, Plaschke CC, Svendsen LB, Gehl J, Achiam MP. Endoscopic electrochemotherapy for esophageal cancer: a phase I clinical study. Endosc Int Open. 2018 Jun;6(6):E727-E734. doi: 10.1055/a-0590-4053. Epub 2018 May 25. PMID 29868638